CLINICAL TRIAL: NCT01886768
Title: Double Versus Single Pledget Method of Nasal Anesthesia for Transnasal Endoscopy: A Randomized Prospective Control Study
Brief Title: Double Versus Single Pledget Nasal Anesthesia for Transnasal Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Chi-Tan Hu, Chief, Division of Gastroenterology, Buddhist Tzu Chi General Hospital, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB101-101
Record Dates: First submitted 2013-02-07; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Anesthesia; Epistaxis
Keywords: Nasal anesthesia; endoscopes; transnasal endoscopy
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double pledget nasal anesthesia (Experimental): All patients in the double pledget nasal anesthesia group receive endoscopic-guided gauze nasal pledgetting to both the inferior nasal meatus and middle nasal meatus. Each patient will receive an anterior rhinoscopy to select the most patent meatus by a validated meatus scoring scale. The endoscope is preloaded with a 1.8 mm biopsy forceps to pick up a right-angled gauze strip. A preloaded biopsy forceps is protruded slowly into the middle meatus first under endoscope monitoring. The second gauze pledgetting procedure is performed two minutes after the first gauze pledgetting which serves to induce turbinate size reduction to both the INT and MNT. A gauze strip is at least brought onto the posterior end of the inferior or middle turbinate.
  Interventions: Device: Double pledget nasal anesthesia (DPNA)
- Single pledget nasal anesthesia (Active Comparator): All patients in the single pledget nasal anesthesia group receive endoscopic-guided gauze nasal pledgetting to either the inferior nasal meatus or middle nasal meatus determined by anterior rhinoscopy. Each patient will receive an anterior rhinoscopy to select the most patent meatus by a validated meatus scoring scale. The endoscope is preloaded with a 1.8 mm biopsy forceps to pick up a right-angled gauze strip. A gauze strip is at least brought onto the posterior end of the inferior or middle turbinate.
  Interventions: Device: Single pledget nasal anesthesia (SPNA)

INTERVENTIONS:
Device: Double pledget nasal anesthesia (DPNA) — By using a transnasal endoscope as a guide and a biopsy forceps, two gauze strips soaked with decongestant and anesthesia will be delivered to the middle meatus followed by the inferior meatus under real-time transnasal endoscopic guidance.
  Other Names: A piece of a 10 X 10 cm Kendall gauze square (Eagle Highland Pharmacy,Indiana, USA) is cut into 4 right-angled triangular gauze strips.; Two right-angled triangular gauze strip are used in DPNA
  Arms: Double pledget nasal anesthesia
Device: Single pledget nasal anesthesia (SPNA) — Another randomized group of patients will also receive endoscopic-guided gauze pledgetting using a transnasal endoscope as a guide and a biopsy forceps. One gauze strip soaked with decongestant and anesthesia will be delivered to either the middle meatus or inferior meatus determined by anterior rhinoscopy.
  Other Names: A piece of a 10 X 10 cm Kendall gauze square (Eagle Highland Pharmacy,Indiana, USA) is cut into 4 right-angled triangular gauze strips.; Only one right-angled triangular gauze strip is used in DPNA.
  Arms: Single pledget nasal anesthesia

SUMMARY:
Unsedated ultrathin transnasal esophago-gastro-duodenoscopy (UT-EGD), in comparison with conventional peroral EGD (P-EGD) has been shown to be more tolerable, safer, cost-effective and time-efficient. The investigators and in other studies have showed that nasal pledgetting (or commonly termed nasal packing) is better than nasal spray in terms of patient tolerance and visual capacity. Although pledgetting method to a selected meatus can achieve better decongestion effect, epistaxis and nasal pain in some patients are still frustrating to endoscopists.

The investigator has proposed a novel meatus scoring scale to evaluate nasal insertability by anterior rhinoscopy using a transnasal endoscope. The investigator also suggest endoscopic-guided gauze pledgetting can provide precise nasal anesthesia, thereby reducing trauma/bleeding in the nasal cavity and increasing patient tolerance during transnasal endoscopy. Endoscopic guidance to deliver a gauze strip can confirm delivering it to at least the posterior end of a turbinate. We hypothesize that by using endoscopic-guided method, gauze pledgetting to both the inferior nasal meatus (INM) and middle nasal meatus (MNM) simultaneously is more tolerable than only gauze pledgetting to a single meatus.

DETAILED DESCRIPTION:
Nasal anesthesia is the rate-limiting step for a well tolerable unsedated transnasal esophago-gastro-duodenoscopy (UT-EGD) procedure. The investigator has proposed that a simple Endoscopic-Guided Gauze Pledgetting method (EGGP) is more tolerable than the "blind" cotton-tippled applicator method to deliver a gauze strip for anesthetizing the nasal cavity. The initial idea of EGGP is to anesthetize only one single selected meatus. To compare patient tolerance, safety and adverse events between double pledget (DPNA, i.e. INM and MNM) versus single pledget (SPNA, i.e. INM or MNM) methods of nasal anesthesia, the investigator is going to conduct a prospective randomized-controlled trial. The rationale for using double pledget is threefold: (1) the middle meatus is bounded by the INT and MNT; (2) the inserting and exserting meatuses may be different; (3) erective spongy tissue is mainly distributed in the inferior and middle turbinates and the nasal septum. Therefore, the primary objective of this study is to evaluate whether DPNA is more tolerable and safer than DPNA before UT-EGD.

ELIGIBILITY:
Inclusion Criteria:

All outpatients with epigastric discomfort (non-ulcer dyspepsia), aged 18-65 years are eligibility for this study.

Exclusion Criteria:

* Patients who can not answer questionnaires, who have prior nasal trauma or surgery, recent or present upper gastrointestinal bleeding and coagulopathy are excluded from this study.
* Patients who are allergic to lidocaine and who have uncontrolled hypertension or coronary artery disease are not recruited.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures are tolerability profiles on a validated visual analogue scale | Immediately after transnasal endoscopy up to all questionnaires answered (about 15 minutes)
  The primary outcome measures are tolerability profiles on a validated visual analogue scale (VAS) and difficulty in inserting the transnasal endoscope through a selected meatus based on a Likert scale. The Likert scale has 5 points of difficulty: minimal, slight, moderate, substantial, and extreme. Facing a 5-point VAS card (1 = minimal discomfort to 5 = severe discomfort), all patients give real-time feedback immediately after UT-EGD by speaking or pointing out their scorings for the following: (1) pain during anesthesia, (2) pain during nasal insertions, (3) pain during exsertion, and (4) overall tolerance.

SECONDARY OUTCOMES:
Secondary outcome measures evaluate the side effects of nasal anesthesia | The immediate secondary outcome measures will be evaluated by questionnaires immediately after UT-EGD within 15 minutes and the delayed secondary outcome measures will be evaluated by otolaryngologists within two weeks after UT-EGD.
  Secondary outcome measures will be evaluated by assisting nurses, who record
  (a) immediate responses including: (i) epistaxis, (ii) immediately post-procedural side effects including headache, light headiness, and mucous discharge, and (iii) patient's willingness to receive the same procedure the next time, and (b) delayed side effect including (i) persisting nasal discharge, (ii) epistaxis 24 hours after UT- EGD, and (iii) sinusitis all confirmed by otolaryngologists within two weeks after UT-EGD. The visual capacity for the anterior nasal cavity ranking on a 5-point scale (5 represented standard EGD and 1 poor visual quality) is also evaluated by assisting nurses during endoscopic insertion after nasal decongestive anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Tan Hu, Principal Investigator — Budhist Tzu Chi Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi Hospital, Hualien City, Hualien county, Taiwan